CLINICAL TRIAL: NCT03162172
Title: Evaluation of the Adult Height Gain With Growth Hormone Treatment in Children With Congenital Adrenal Hyperplasia (CDAH), Using the OPALE Prediction Model
Brief Title: Growth Hormone (GH) in Congenital Adrenal Hyperplasia
Acronym: OPALE GH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CIC 2009-019
Record Dates: First submitted 2017-05-16; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Adrenal Hyperplasia, Congenital
Keywords: congenital adrenal hyperplasia; short stature; growth hormone treatment
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Dwarfism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital adrenal hyperplasia (CAH) is a genetic rare disease, which alters the adrenal production of gluco and mineralo corticoids. The treatment consists in supplementing children using hydrocortisone. Despite care for these children has improve substantially across decades, short adult height still remains an important consequence of the disease. About 20 % of patients have an AH below 2 standard deviations compared to their expected height.

In the OPALE model study, the investigators have collected data from a cohort of 496 French patients, born between 1970 and 1991 and with a known genotype. Using their age, sex, growth, disease, bone maturation and pubertal data, they have built a model which allows to predict their AH using data available at 8 years of age. This model has shown that the currently used formula to calculate the predicted AH (Bayley Pineau's method) is not applicable to children with CAH.

In this project, the investigators plan to use the prediction model to compare the AH in patients who have received GH treatment to their predicted AH using the model.

The hypothesis is that GH improves the AH in such patients. Existing cohorts have shown improved growth celerity, and growth expectation using the Bayley-Pineau formula), but this has not been shown on the actual AH.

This study will allow to reinforce the investigators' hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Patients with CAH, born between 1970 and 1998, having received GH treatment for a minimal one year duration.

Exclusion Criteria:

* Patients with chronic any growth altering disease, Turner syndrome or other genetic anomaly; 8-year wrist Xray and adult height should be available to allow the use of the OPALE model prediction.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with genetically proven CAH, classical form, or simple virilizing, with 21 hydroxylase, or 11ᵝ hydroxylase, or 3βol-dehydrogenase deficit, born between 1970 and 1998, having received GH treatment for a minimal one year duration.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
Adult height (AH) gain | up to 18 years
  Difference between AH predicted by the OPALE model, and observed AH defined as (i) the height recorded after age 20 in boys or 18 in girls; (ii) the height recorded when bone age (BA) is ≥ 18 years in boys and 16 years in girls (99.6% of AH) (10); or (iii) the height measured after growth velocity drop to ≤ 1 cm/year

SECONDARY OUTCOMES:
Number of treatment withdrawal due to adverse events | up to 6 years of GH treatment
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bretones, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No